CLINICAL TRIAL: NCT00293085
Title: An Open, Randomized, Multicentre, Phase II Pilot Study of Docetaxel and Cisplatin in the Adjuvant Treatment of Non-Small Cell Lung Cancer (NSCLC) Stage I-II
Brief Title: An Open, Randomized, Multicentre, Phase II Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Prof. Dr. Thomas Brodowicz, CECOG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/ NSCLC 2.2.001
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Active Comparator): Docetaxel (Taxotere ) 75 mg/m² as a 1 hour i.v. infusion, followed immediately by cisplatin 75 mg/m² as a 1 hour i.v. infusion, on day 1 every 21 days for 6 cycles.
  Dose reductions and/or treatment delays or discontinuation of treatment are planned for arm A in case of severe haematological and/or non haematological toxicities.
  Premedication:
  Dexamethasone 8 mg p.o. (or any other steroid commonly used) will be given -12 h, -3 h, -1 h before start of docetaxel infusion, then + 12 h, +24 h and + 36 h post infusion.
  All patients should receive a prophylactic antiemetic premedication to prevent nausea and vomitus, which includes a 5-HT3 antagonist prior to start of each docetaxel infusion.
  Hyperhydration Patients will require intravenous hydration according to institutional guidelines.
  Interventions: Drug: Docetaxel
- Comparative arm (No Intervention): No chemotherapy will be administered. No specific salvage therapy after progression is defined.

INTERVENTIONS:
Drug: Docetaxel
  Arms: Docetaxel
Drug: Docetaxel — Docetaxel (Taxotere) 75 mg/m² as a 1 hour i.v. infusion, followed immediately by cisplatin 75 mg/m² as a 1 hour i.v. infusion, on day 1 every 21 days for 6 cycles.
  Dose reductions and/or treatment delays or discontinuation of treatment are planned for arm A in case of severe haematological and/or non haematological toxicities.
  Premedication:
  Dexamethasone 8 mg p.o. (or any other steroid commonly used) will be given -12 h, -3 h, -1 h before start of docetaxel infusion, then + 12 h, +24 h and + 36 h post infusion.
  All patients should receive a prophylactic antiemetic premedication to prevent nausea and vomitus, which includes a 5-HT3 antagonist prior to start of each docetaxel infusion.
  Hyperhydration Patients will require intravenous hydration according to institutional guidelines.
  Arms: Docetaxel

SUMMARY:
The objective of this study is to evaluate efficacy, safety and quality of life adjuvant docetaxel-cisplatin chemotherapy versus no adjuvant treatment in patients with completely resected NSCLC Stage I-II.

DETAILED DESCRIPTION:
Open multicentre, centrally randomized, two-arm parallel-group, phase II pilot-study. Duration of the Treatment : Arm A - will be 4-6 cycles Docetaxel 75mg/m2 and Cisplatin 75mg/m2 on day 1 every 21 days.

Arm B untreated control group - best supportive care. A follow-up check-up examination will be performed every 3 months for a total of three years.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented NSCLC stage I-II
* Complete resection of tumor amd resection margins microscopically tumor free.
* Surgical procedure: According to necessity for oncology radicality a lobectomy, bilobectomy or pneumectomy will be performed with either radical mediastinal lymphadenectomy or complete sampling of all relevant lymph node areas.
* Randomization within 60 days after surgical required.
* Initial work-up
* General Conditions: 19-70 years, WHO performance status 0-2, adequate hematological function, adequate renal and hepatic function, negative pregnancy test.

Exclusion Criteria:

* NSCLC stage II-IV, SCLC or alveolar carcinoma
* Clinical evidence of CNS metastases
* pregnant and lactating patients
* past or concurrent history of malignancies other than NSCLC,except for curatively treated non melanoma of the skin or in situ cervical carcinoma or other curatively treated cancer with no evidence of disease for at least five years.
* prior or concurrent antitumor therapy for NSCLC other than surgery.
* Concomitant participation in clinical studies of non-approved experimental agents or procedures.
* major complications after surgery
* serious concomitant medical conditions
* psychological,familial, sociological or geographical conditions which do not permit compliance with the study protocol

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2001-12; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
to compare the effect on disease free survival of adjuvant docetaxel and cisplatin in patients with completely resected stage I-II non-small cell lung cancer versus observation only

SECONDARY OUTCOMES:
to determine the impact on overall survival of adjuvant docetaxel and cisplatin.
to characterise and quantitate toxicity related to this treatment regimen.
to compare quality of life of patients on both treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph C. Zielinski, Prof, Principal Investigator — Univ. Klinik f. Innere Medizin I

REFERENCES:
- See also: Related Info — http://www.cecog.org